CLINICAL TRIAL: NCT01582048
Title: Multicenter Phase II Study of Peritransplantation Immunosuppression Using ATG, Rituximab, Sirolimus and Mycophenolate Mofetil in Patient Receiving Mismatched Hematopoietic Cell Transplantation After Reduced Intensity Conditioning With Fludarabine and Treosulfan
Brief Title: Multicenter Study of Peritransplantation Immunosuppression for Mismatched Hematopoietic Cell Transplantation After Reduced Intensity Conditioning
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Prof. Dr. med. Wolfgang Bethge (Other)
Collaborators: medac GmbH (Industry); Pfizer (Industry); Neovii Biotech (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Wolfgang Bethge, Associate Professor Hematology/Oncology, University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E:531/2011; 2011-002192-41 (EudraCT Number)
Record Dates: First submitted 2012-04-16; First posted 2012-04-20 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Patients Receiving Mismatched Allogeneic HCT
MeSH Terms: interventions — Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: immunosuppression — Conditioning with treosulfan 14 g/m2 day -6 to -4, fludarabine 30 mg/m2/24h day-6 to -2, ATG-Fresenius 20 mg/kg day -4 to -2, rituximab 500 mg/m2 day -1. Unmanipulated PBSC day 0. Postgrafting immunosuppression with mycophenolate mofetil (15 mg/kg TID) and sirolimus (2 mg QD).

SUMMARY:
Feasibility and toxicity of peritransplantation immunosuppression with ATG, sirolimus, mycophenolate mofetil and rituximab in patients receiving mismatched allogeneic HCT after a reduced intensity conditioning regimen with fludarabine/treosulfan

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for mismatched allogeneic HCT
* Unrelated donor with maximal 2 antigen or allelic mismatches in HLA-I or HLA-II
* Age >=75, >=18 years
* Patients Age <=50 if a HCT-CI score > 2 [acc. to Sorror et al., 2005]
* Karnofsky Index >60%
* Patients with:

  * Acute myeloid leukemia in CR (<5% blasts)
  * Acute lymphoblastic leukemia in CR (< 5% blasts)
  * Myelodysplastic syndrome with up to 20% blasts
  * Osteomyelofibrosis
  * Chronic lymphocytic leukemia
  * High grade Non-Hodgkin Lymphoma in CR or PR
  * Low grad Non-Hodgkin Lymphoma in CR or PR
  * M. Hodgkin in CR or PR
  * Chronic myeloid leukaemia in chronic phase or CR of blast crisis

Exclusion Criteria:

* Patients with >5% blasts in BM at the time of transplantation
* Progressive or chemorefractory disease
* Less than 3 months after preceding HCT
* CNS involvement with disease
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month.
* Liver function abnormalities with bilirubin >2 mg/dL and elevation of transaminases higher 2x upper limit of normal.
* Chronic active viral hepatitis
* Ejection fraction <40 % on echocardiography
* Patients with > grade II hypertension by CTC criteria
* Creatinine clearance <50 ml/min
* Proteinuria >800 mg/24 h
* Respiratory failure necessitating supplemental oxygen or DLCO <30%
* Allergy against murine antibodies
* Known allergy/intolerance against sirolimus or one of it's excipients
* HIV-Infection
* Female patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control during study treatment and for at least 12 months thereafter. (Women of childbearing potential must have a negative serum pregnancy test at study entry)
* Concurrent severe and/or uncontrolled medical disease (e.g. uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months prior to the study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study
* Patients with a history of psychiatric illness or condition which could interfere with their ability to understand the requirements of the study (this includes alcoholism/drug addiction)
* Patients unwilling or unable to comply with the protocol
* Unable to give informed consent
* Enrollment in an other trial interfering with the endpoints of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-04; Primary Completion 2016-08-17 (Actual); Study Completion 2016-08-17 (Actual)

PRIMARY OUTCOMES:
Treatment related mortality | 12 months after HCT
Treatment related mortality | 24 months after HCT

SECONDARY OUTCOMES:
Toxicity according CTC of protocol on day 100 | on day 100
Engraftment on day 100 | on day 100
Overall survival | 12 months after HCT
Incidence of graft versus host disease | 3 months after HCT
Incidence of infections | 2 years after HCT
Immune reconstitution of CD3, CD3/CD4/CD8, CD56, CD19 cells | 3 months after HCT
Overall survival | 24 months after HCT
Incidence of graft versus host disease | 6 months after HCT
Disease free survival | 24 months after HCT
Disease response | 12 months after HCT
Disease response | 24 months after HCT
Immune reconstitution of CD3, CD3/CD4/CD8, CD56, CD19 cells | 6 months after HCT
Immune reconstitution of CD3, CD3/CD4/CD8, CD56, CD19 cells | 12 months after HCT
Immune reconstitution of CD3, CD3/CD4/CD8, CD56, CD19 cells | 24 months after HCT
Incidence of graft versus host disease | 12 months after HCT
Incidence of graft versus host disease | 24 months after HCT

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang A Bethge, MD, Principal Investigator — Medical Center University Hospital of Tuebingen
Locations (4):
- Germany (4):
  - Hematology/Oncology Medical Center University Hospital of Mainz, Mainz
  - Bone Marrow Transplantation Unit Medical Center University Hospital of Nuernberg, Nuremberg
  - Department of Hematology/Oncology Medical Center University Hospital of Tuebingen, Tübingen
  - BMT-Unit Deutsche Klinik für Diagnostik, Wiesbaden

REFERENCES:
- See also: Results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2011-002192-41